CLINICAL TRIAL: NCT01205087
Title: Safety and Efficacy of Oral Administration of Anti-CD3 Monoclonal Antibody in Patients With the Metabolic Syndrome PHASE IIa A Single-blinded Placebo-controlled Clinical Trial
Brief Title: Safety and Efficacy of Oral Administration of Anti-CD3 Monoclonal Antibody (mAb)in Patients With the Metabolic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Collaborators: NasVax Ltd (Industry)
Responsible Party: Gadi Lalazar, M.D., Department of Medicine, Hadassah University Hospital, Jerusalem, Israel
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OKT3-NASH-HMO-CTIL
Record Dates: First submitted 2010-05-23; First posted 2010-09-20 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Muromonab-CD3; Omeprazole

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: OKT3
- OKT3 - 0.2 (Active Comparator)
  Interventions: Drug: OKT3
- OKT3 - 1 (Active Comparator)
  Interventions: Drug: OKT3
- OKT3 - 5 (Active Comparator)
  Interventions: Drug: OKT3

INTERVENTIONS:
Drug: OKT3 — Oral anti-CD3 MAb will be administered at a dosage level of 0.2 or 1.0 or 5.0 mg per day for 30 days. Up of 9 patients will be treated at each dosage level, and up to additional 9 patients will receive placebo.
  Other Names: Omeprazole

SUMMARY:
This clinical study is designed to evaluate the safety and immune modulatory effects of oral administration of the study drug anti-CD3 monoclonal antibody (MAb) to subjects with the metabolic syndrome.

DETAILED DESCRIPTION:
PHASE IIa STUDY PROTOCOL A Single-blinded Placebo-controlled Clinical Trial.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who have completed the informed consent process culminating with written informed consent by the subject.
2. Men and women age 18 to 75 years (inclusive)
3. Patients with biopsy proven NASH within the last 3 years
4. Altered glucose metabolism, including diabetes (non treated, or treated with up to 2 drugs (not including insulin) without any change in medication for at least 2 months prior to enrollment), impaired fasting glucose or impaired glucose tolerance.
5. HBA1C between 5.5 and 14%.

Exclusion Criteria:

1. Subjects who have undergone surgery within the last 3 months.
2. Subjects who have had a prior gastrointestinal surgery.
3. Subjects with a clinically significant infectious, immune mediated or malignant disease
4. Subjects who are receiving an elemental diet or parenteral nutrition.
5. Subjects who have been treated with any type of immune modulatory drug including steroids or NSAID within the last 4 weeks
6. Subjects who have received either methotrexate or cyclosporine or anti TNF-β (infliximab, Remicade), anti-integrin (namixilab) or who have participated in any other clinical trial within the last 3 months.
7. Subjects with a history of coagulopathy.
8. Women with childbearing potential unless surgically sterile or using adequate contraception (either IUD, oral or Depo-provera contraceptive, or barrier plus spermicide); pregnant or breastfeeding mothers.
9. Subjects, who will be unavailable for the duration of the trial, are unlikely to be compliant with the protocol, or who are felt to be unsuitable by the investigator for any other reason.
10. Subjects who are HIV-positive.
11. Subjects who are HBV-positive
12. Subjects who are HCV-positive.
13. Subjects with active CMV
14. Subjects with anemia (Hb <10.5 gm/dl).
15. Subjects with thrombocytopenia (platelets <100K/µl).
16. Subjects with lymphopenia (absolute lymphocyte count <0.7).
17. Subjects with IgG anti-cardiolipin antibody >16 IU.
18. Prior exposure to anti-CD3 MAb.
19. Known sensitivity to any ingredients in the study drug
20. Any know autoimmune disease except for the studied disorders.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2010-09; Primary Completion 2010-12 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
This clinical study is designed to evaluate the safety and the immune-modulatory effects of oral administration of the study drug anti-CD3 MAb to subjects with the metabolic syndrome. | 60 days

SECONDARY OUTCOMES:
This clinical study also will include evaluations for markers of efficacy, as described below. | 60 days

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah University Hospital, Liver Unit, Jerusalem, Israel